CLINICAL TRIAL: NCT01700270
Title: A Phase I, Multi-center, Open-label, Drug-drug Interaction Study to Assess the Effect of the CYP1A2 Inhibitor, Fluvoxamine, on Dovitinib (TKI258) Pharmacokinetics in Patients With Advanced Solid Tumors
Brief Title: Pharmacokinetic Drug-drug Interaction Study of Dovitinib (TKI258) in Patients With Advanced Solid Tumors.
Acronym: CTKI258A2120
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2120; 2012-001546-18 (EudraCT Number)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2014-11

CONDITIONS: Advanced Solid Tumors, Excluding Breast Cancer
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Fluvoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dovitinib (TKI258) (Experimental): dovitinib, 5 days on / 2 days off dose schedule
  Interventions: Drug: dovitinib (TKI258); Drug: fluvoxamine

INTERVENTIONS:
Drug: dovitinib (TKI258)
Drug: fluvoxamine — perpetrator drug; 7 days of dosing

SUMMARY:
This is a multi-center, open-label, single-sequence, crossover, drug-drug interaction (DDI) study to assess the effect of the CYP1A2 inhibitor, fluvoxamine, on the PK of dovitinib in patients with advanced solid tumors, excluding breast cancer. The purpose of this study is to evaluate the effect of a CYP1A2 inhibitor, 100 mg fluvoxamine, on the PK of dovitinib when administered at a dose of 300 mg on the dosing schedule, 5 days on/2 days off. The study will consist of 2 phases: a Pharmacokinetic (PK) phase and a clinical treatment phase. The DDI test will be conducted in the PK phase. The DDI test will assess the steady state PK profile of dovitinib when administered alone and in the presence of the CYP1A2 inhibitor, fluvoxamine (AUC 0-24h, AUC 0-72h and Cmax parameters). During the clinical treatment phase patients may continue to receive treatment with TKI258 until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death or discontinuation from the study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

Patients with a cytopathologically or histopathologically confirmed diagnosis of an advanced solid tumor, excluding breast cancer which has progressed despite standard therapy or for which no standard therapy exists - ECOG performance status 0 or 1 and an anticipated life expectancy of ≥3 months- Patient must meet protocol-specific laboratory values

Exclusion Criteria:

- Patients with brain metastases - Patients who have received or who are expected to receive any prohibited medications and therapies - Patients who have received CYP1A2 or CYP3A inhibitor medications within 5 days prior to start study treatment or are expected to receive during the first 28 days after starting the study treatment - Patients who have received CYP1A2 or CYP3A inducer medications within 30 days prior to start study treatment or are expected to receive during the first 28 days after starting the study treatment - Patients who are actively taking antidepressants, benzodiazepines, serotonergic drugs, and/or monoamine oxidase inhibitors (MAOIs) - Patients who have not recovered from previous anti-cancer therapies - Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of TKI258 - Patients who have concurrent severe and/or uncontrolled concomitant medical conditions that could compromise participation in the study - Female patients who are pregnant or breast-feeding - Fertile males or women not willing to use highly effective methods of contraception - Other protocol-defined inclusion/exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
TKI258 pharmacokinetics (PK) parameters: Cmax (Maximum (peak) concentration of drug) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: AUC 0-24 hr (Area Under the Curve) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: AUC 0-72 hr | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: Tmax (Time to maximum concentration) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: T1/2 (Half-life time) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: CL/F (Apparent Oral Clearance) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)
TKI258 pharmacokinetics (PK) parameters: Vz/F (apparent volume of distribution) | multiple time-points over 72h post dose on day Day 19 and Day 26 (PK phase)

SECONDARY OUTCOMES:
Frequency and severity of AEs (Adverse Events) | up to at least 30 days after the last dose of dovitinib (TKI258)
Frequency and severity of SAEs (Serious Adverse Events) | up to at least 30 days after the last dose of dovitinib (TKI258)
Preliminary evidence of antitumor activity of dovitinib (TKI258) | every 8 weeks until progression of disease
  overall response based on investigator assessment and best overall response using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (2):
  - Montefiore Medical Center Montefiore Medical Center (SC), The Bronx, New York
  - Cancer Therapy & Research Center / UT Health Science Center SC, San Antonio, Texas
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Amsterdam, Netherlands
- Switzerland (2):
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Geneva

REFERENCES:
- [Derived] de Weger VA, Goel S, von Moos R, Schellens JHM, Mach N, Tan E, Anand S, Scott JW, Lassen U. A drug-drug interaction study to assess the effect of the CYP1A2 inhibitor fluvoxamine on the pharmacokinetics of dovitinib (TKI258) in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2018 Jan;81(1):73-80. doi: 10.1007/s00280-017-3469-4. Epub 2017 Nov 3. PMID 29101463
- See also: Results for CTKI258A2120 on the Novartis Clinical Trial Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13925